CLINICAL TRIAL: NCT04400370
Title: Point of Care Ultrasound to Evaluate Diaphragmatic Function in Children Undergoing Thoracic Surgery: Prospective Observational Study
Brief Title: Point of Care Ultrasound to Evaluate Diaphragmatic Function in Children Undergoing Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: diaphragm_US
Record Dates: First submitted 2020-05-06; First posted 2020-05-22 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Diaphragm Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients undergoing lung resection
  Interventions: Device: Diaphragm ultrasound

INTERVENTIONS:
Device: Diaphragm ultrasound — Diaphragm ultrasound is performed at the following three time points.
  1. At the entrance of the operating room before induction of anesthesia
  2. 1 hour after surgery
  3. 24 hours after surgery

SUMMARY:
In children undergoing pulmonary resection, the diaphragm function is evaluated using ultrasound before and after surgery to evaluate the incidence of diaphragm dysfunction after pulmonary resection. In addition, we examine if there is a relationship between diaphragmatic dysfunction and pulmonary complications, including postoperative lung atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under 7 years undergoing lung resection

Exclusion Criteria:

* Asthma
* Myopathy or neuropathy

Max Age: 6 Years | Sex: All
Age Groups: Child
Study Population: Pediatric patients under 7 years undergoing lung resection
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in diaphragmatic thickness | 1. Before the procedure; 2. 1 hour after surgery; 3. 24 hours after surgery
  Changes in diaphragmatic thickness, from time frame 1 to 3
Changes in diaphragm thickening fraction | 1. Before the procedure; 2. 1 hour after surgery; 3. 24 hours after surgery
  Changes in diaphragm thickening fraction, from time frame 1 to 3
Changes in the length of diaphragmatic tidal excursion | 1. Before the procedure; 2. 1 hour after surgery; 3. 24 hours after surgery
  Changes in the length of diaphragmatic tidal excursion, from time frame 1 to 3

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Kang P, Park JB, Kim JT. Changes in diaphragmatic ultrasonography findings and their association with postoperative complications in children undergoing pulmonary resection: A single-centre, prospective, observational study. Eur J Anaesthesiol. 2023 Dec 1;40(12):953-956. doi: 10.1097/EJA.0000000000001910. Epub 2023 Oct 12. PMID 37823729